CLINICAL TRIAL: NCT03779256
Title: ENDO - Bowel ENDOmetriosis; Evaluation of Diagnostics and Quality of Life (ENDO1, ENDO2, ENDO3)
Brief Title: Bowel ENDOmetriosis; Evaluation of Diagnostics and Quality of Life
Acronym: ENDO
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: St John of God Hospital, Vienna (Other); Nepean Blue Mountains Local Health District (Other)
Responsible Party: Principal Investigator, Kristine Aas-Eng, Principal investigator, Oslo University Hospital
Other Study IDs: 2017/1925 REK Sør-Øst D
Record Dates: First submitted 2018-12-04; First posted 2018-12-19 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Endometriosis Related Pain; Quality of Life; Pain, Chronic; Bowel Dysfunction; Endometriosis Rectum; Deep Infiltrating Endometriosis; Deep Endometriosis
Keywords: Deep infiltrating endometriosis; Transvaginal ultrasound; Endometriosis rectum; Conservative surgery; Radical surgery; Quality of life; Deep endometriosis
MeSH Terms: conditions — Chronic Pain; Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bowel excised by discoid excision or segmental resection sent for histopathological examination, which is routine practice after surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with bowel endometriosis.: Women with symptomatic bowel endometriosis scheduled for surgical treatment investigated with 2D transvaginal ultrasound before surgery at Hospital St John of God, Vienna, Austria; Oslo university hospital, Oslo, Norway and Nepean Hospital, Sydney, Australia.
  The women recruited at Oslo university hospital, Norway will also have a magnetic resonance imaging (MRI) of the abdomen and pelvis before surger.
  Interventions: Procedure: 2D transvaginal ultrasound

INTERVENTIONS:
Procedure: 2D transvaginal ultrasound — Transvaginal ultrasound is part of routine pre-operative examination of the women before surgery is scheduled. Described surgical treatment interventions is standard practice used to alleviate patient symptoms.
  Women recruited at Oslo university hospital, Norway will also have an MRI performed pre-operatively.
  Other Names: Segmental bowel resection or; Disc excision of bowel

SUMMARY:
Endometriosis on the bowel is a benign condition that can cause major complaints and severely affect the quality of life of women of fertile age. If medical treatment is not enough to improve pain and/or other symptoms it may be necessary to undergo major surgical treatment and removal of the endometriosis nodule on the bowel. Such extensive surgical treatment carries risks of serious complications. Therefore, a thorough diagnostic work-up before surgery is important to know the extent of disease. This will provide women with the best possible information and for the surgeon to plan the operation. The risk of complications increases as the bowel endometriosis is localized closer to the anus as well and/or if the bowel nodule is large.

The distance between the anus and the nodule and the size of the nodule can be measured with two dimensional (2D) vaginal ultrasound. Additionally, Magnetic resonance imaging (MRI) is also used in some countries for these same measurements. Our study would like to investigate the diagnostic value of 2D ultrasound and MRI as well as learn more about women's quality of life before and after surgery. The investigators have designed the study to evaluate the following three questions into three studies ENDO1, ENDO2 and ENDO3:

* ENDO1: How good is 2D transvaginal ultrasound at measuring the size of the bowel endometriosis nodule and the distance between anus and the lower part of the bowel nodule compared to measurements done during surgery?
* ENDO2: What is the quality of life, sexual and bowel function of women before and 3- and 12-months after surgery due to bowel endometriosis? Questionnaires will be used.
* ENDO3: How good is 2D transvaginal ultrasound at measuring the size of the bowel endometriosis nodule compared to magnetic resonance imaging (MRI) and measurements done during surgery?

DETAILED DESCRIPTION:
Mild endometriosis normally affects the peritoneum. More advanced form of endometriosis is termed deep infiltrating endometriosis (DIE). In women suffering from DIE, the endometriotic tissue invades the tissue >5mm below the peritoneal surface, affecting organs in the pelvis like the ovaries, uterus, vagina, bladder, ureters and/or bowel. In women with suspected endometriosis, the prevalence of DIE affecting the bowel is found to range from 24.0 to 73.3%. The symptoms of DIE can be debilitating with dysmenorrhoea, dyspareunia, altered bowel motions, dyschezia and/or dysuria. Thus, it may have an immense impact on women's quality of life with societal consequences.

The risk of complications with surgery for deep infiltrating endometriosis (DIE) of the bowel can be severe like anastomotic leak and rectovaginal fistula. Evidence show that there is an increased risk of anastomotic leaks bowel if the anastomosis <5-8cm from the anal verge. DIE of the rectosigmoid colon can be diagnosed by widely available and low-cost two-dimensional transvaginal sonograhpy (2D-TVS) with a high sensitivity and specificity. MRI is comparable to TVS in diagnosis of intestinal endometriosis but is costlier and less available than TVS. MRI has the advantage over 2D-TVS that it is reproducible, the area of interest can be viewed in many planes and the images can be reviewed and compared by same or different examiners over time.

There are two surgical approaches used in women suffering from bowel endometriosis, namely segmental resection of rectosigmoid or nodule excision. Nodule excision may be performed by shaving (not opening the rectum) or disc excision (removing bowel nodule with surrounding rectal wall). The success of pelvic pain reduction following surgery in women suffering from DIE is related to the radicality of surgery. However, some argue a more symptom-guided approach to surgery.

Endometriosis itself and surgical treatment may have immense impact endometriosis can have on a woman's life. Thus, it is essential to discuss the severity of symptoms, any implications of surgery as well as the risk of complications to enable women informed consent. The pre-operative information and decision making is based on symptoms, fertility wish, the clinical examination and diagnostic tests. Consequently, diagnostic tools such as TVS and MRI are important factors to plan and perform a safe procedure with the best possible outcomes for the women.

There are, to the investigator's knowledge, no studies, which demonstrate if there is a correlation between measurement of the size of an endometriotic rectosigmoid lesion with 2D-TVS compared to the actual lesion size in the resected bowel. Additionally, there are no studies that investigate the correlation between the distance between the rectosigmoid lesion and the anal verge, to plan appropriate surgery and estimate risk of serious complications. Furthermore, there are no known studies evaluating the correlation of measurements of bowel lesions when comparing transvaginal 2D-TVS, MRI and surgery. The aim of surgery is to improve women's quality of life and thus it is essential to evaluate results before and after surgery for bowel endometriosis.

ELIGIBILITY:
Inclusion Criteria:

- Women of reproductive age, ≥ 18 years old, scheduled for planned laparoscopic or open bowel surgery for deep infiltrating endometriosis with suspected symptomatic bowel lesions.

Exclusion Criteria:

- Postmenopausal women, women < 18 years old, women with previous bowel surgery. Women who do not speak and read fluent English or Norwegian.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Eligible women will be included from tertiary referral centers for deep infiltrating endometriosis.
  ENDO1 will include women from Oslo University Hospital, Hospital St John of God and Nepean Hospital. Estimated total eligible women: 135.
  ENDO2 will include women from Oslo University Hospital and Nepean Hospital. Estimated eligible women: 70.
  ENDO3 will include women from Oslo University Hospital. Estimated eligible women: 40
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
ENDO1AMeasurements on the distance between the lower margin of the rectal lesion and anal verge with 2D-TVS | Before scheduled surgery
  Millimeter distance measured on 2D TVS
ENDO1A: Measurements on the distance between the lower margin of the rectal lesion and anal verge | During scheduled surgery
  Millimeter distance measured during surgery
ENDO1B: Size of bowel lesion measured on the excised bowel lesion. | During surgery.
  Millimeter measurements of the bowel lesion in three orthogonal planes i.e. mid-sagittal, anteroposterior and transverse according to the IDEA group.
ENDO1B: Size of bowel lesion measured with 2D-TVS. | Before scheduled surgery.
  Millimeter measurements of the bowel lesion in three orthogonal planes i.e. mid-sagittal, anteroposterior and transverse according to the IDEA group.
ENDO2: Incidence of low anterior resection syndrome (LARS) | Preoperatively, 3- and 12-months postoperatively
  LARS questionnaire consisting of five questions, each response correlates to a score. Lowest score is 0-20 i.e. no LARS, score 21-29 i.e. minor LARS and score 30-42 i.e. major LARS.
ENDO3: Correlation between Lesion to anal verge distance (LAVD) measured with 2D-TVS, MRI and measurements during surgery | Pre-operatively and during surgery
  Millimeters of lesion to anal verge distance measured
ENDO3: Measurements of bowel lesion size with MRI compared to 2D TVS and surgery | Before and during scheduled surgery
  Millimeter measurements of the bowel lesion in three orthogonal planes i.e. mid-sagittal, anteroposterior and transverse according to the IDEA group.

SECONDARY OUTCOMES:
ENDO1: Numerical analogue scale (NAS) score of dysmenorrhea, dyspareunia, dyschezia, dysuria. | Preoperatively, 3 and 12 months postoperatively
  Numerical analogue scale ranging from 0 to 10 scored for each symptom, 0 representing no pain and 10 representing worst possible pain
ENDO1: Type and frequency of complications after bowel surgery | Through study completion, an average of 1 year
  "Clavien-Dindo" classification of surgical complications
ENDO2: Quality of life Endometriosis Health Profile-30 | Preoperatively, 3 and 12 months postoperatively
  Using questionnaire - Endometriosis Health Profile (EHP-30), consisting of a core questionnaire with 30 items grouped into 5 scales and modular questionnaire consisting of 23 items grouped into 6 scales. All scales have a minimum score of 0 (indicating low disability) and a maximum score of 100 (indicating high disability).
ENDO2: Sexual function | Preoperatively, 3 and 12 months postoperatively
  Using questionnaire - Female Sexual Function Index (FSFI) consisting of 19 questions, minimum score 2.0 (worst score), maximum score 36.0 (best score).
ENDO2: Quality of life before bowel surgery | Before surgery
  GIQLI (gastrointestinal quality of life index) questionnaire. 36 questions, each containing 4 answers equating to a score ranging from 0 (least desirable answer) to 4 (most desirable answer). Total score range 0-144.
ENDO2: Quality of life after bowel surgery | 3 months
  GIQLI questionnaire
ENDO2: Quality of life after bowel surgery | 12 months
  GIQLI questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mee Kristine Aas-Eng, MD, Principal Investigator — Oslo University Hospital
Locations (3):
- Nepean Hospital, Sydney, Australia
- Hospital St John of God, Vienna, Austria
- Oslo university hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided